CLINICAL TRIAL: NCT00632528
Title: Evaluation of the Efficacy of "MEOPA" Used to Obtain Better ROM Immediately After Multilevel Surgery in Children With Spastic Diplegia, Quadriplegia or Hemiplegia.
Brief Title: MEOPA to Improve Physical Therapy Results After Multilevel Surgery
Acronym: KINOPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P061007; CRC 06 013 (Other: CRC)
Record Dates: First submitted 2008-02-28; First posted 2008-03-10 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2008-02

CONDITIONS: Cerebral Palsy; Spastic Diplegia; Quadriplegia; Hemiplegia
Keywords: MEOPA; spasticity; multilevel surgery; cerebral palsy; children
MeSH Terms: conditions — Cerebral Palsy; Quadriplegia; Hemiplegia; Muscle Spasticity | interventions — Meopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Administration of MEOPA gaz during postoperative physical therapy
  Interventions: Drug: MEOPA
- 2 (Placebo Comparator): Administration of medical air during postoperative physical therapy
  Interventions: Drug: Medicinal air

INTERVENTIONS:
Drug: MEOPA — Administration of MEOPA gaz during postoperative physical therapy
  Arms: 1
Drug: Medicinal air — Administration of medical air during postoperative physical therapy
  Arms: 2

SUMMARY:
Children with cerebral palsy commonly undergo "multilevel surgery", meaning several lower limb combined procedures performed during the same surgical intervention. The aim of this type of surgery is to correct all deformities together in order to restore near to normal anatomy and muscular function. It is very important to be able to obtain good range of motion after surgery, in order to consolidate surgical results. During the first days after the operation, children are sore and it may be difficult to realize adequate physical therapy. In order to palliate this situation, MEOPA gaz is used during REHAB sessions. Good results have been obtained so far but no study is available to demonstrate these results. The goal of our research is to prove that there is a benefit in using MEOPA postoperatively in these patients.

DETAILED DESCRIPTION:
The study is a randomized, single blinded, controlled clinical trial. It consist of two groups of patients: one group will receive MEOPA (FDA approval-"AMM" in France, 2003) and the other will receive medical air.

Results, in terms of articular range of motion, will be compared between groups after five sessions of REHAB. The following items will be evaluated: degree of pain, measured by a pain scale; joint ROM; number of sessions to obtain the desired results; parents, patients and caregivers satisfaction.

Patients aging from 6 to 20 years will be included if they meet selection criteria. Inclusions are confirmed before the first session starts. At this time, informed consent is to be signed by patients or parents and the Clinical Epidemiology Unit will assign a study number to the patient.

All patients get morphine therapy before the REHAB session; a new dose is administrated 10 minutes later if pain is higher than 4/10; ten minutes later, if pain is still over 4/10, MEOPA (or medical air) will be administrated. If this is not enough to diminish pain, the session will be interrupted. Five physical therapy sessions are provided after surgery, during inpatient time.

Knee ROM will be measured by goniometry and will be the measure of reference to evaluate the influence of MEOPA. Two types of pain scale will be used: analogical scale from 1 to 10 and faces scale (FPS-R) for small children.

For security reasons, the person who administrates de gaz will be informed of the nature of the product (MEOPA or medical air), the bottle will be masked and the therapist won't know what kind of product is being administrated.

ELIGIBILITY:
Inclusion Criteria:

* Multilevel surgery
* Spastic cerebral palsy

Exclusion Criteria:

* Patient not being able to walk

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Knee range of motion | at 7 days

SECONDARY OUTCOMES:
Improvement of function after surgery | at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ana PRESEDO, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré University Hospital, Paris, France

REFERENCES:
- [Result] Delafontaine A, Presedo A, Mohamed D, Lopes D, Wood C, Alberti C. Equimolar mixture of nitroux oxyde and oxygen during post-operative physiotherapy in patients with cerebral palsy: A randomized, double-blind, placebo-controlled study. Eur J Pain. 2017 Nov;21(10):1657-1667. doi: 10.1002/ejp.1071. Epub 2017 Jul 20. PMID 28726270